CLINICAL TRIAL: NCT05126667
Title: A Propensity Score-Matched Analysis of Breast-Conserving Surgery Plus Whole-Breast Irradiation Versus Mastectomy in Breast Cancer
Brief Title: Analysis of Breast-Conserving Surgery Plus Whole-Breast Irradiation Versus Mastectomy
Status: Completed | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID 2762
Record Dates: First submitted 2021-11-17; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental; Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast-conserving surgery: Patients who underwent breast-conserving surgery plus whole-breast irradiation
  Interventions: Procedure: Breast-conserving surgery
- Mastectomy: Patients who underwent mastectomy
  Interventions: Procedure: Mastectomy

INTERVENTIONS:
Procedure: Breast-conserving surgery — Breast conserving surgery plus whole breast irradiation
  Groups: Breast-conserving surgery
Procedure: Mastectomy — Breast mastectomy
  Groups: Mastectomy

SUMMARY:
This is a retrospective propensity score-matched analysis of a large institutional cohort of patients in order to compare long-term outcomes and clinicopathologic characteristics between patients treated with breast conserving surgery or mastectomy for breast cancer.

DETAILED DESCRIPTION:
The aim of the study is to compare long-term outcomes and clinicopathologic characteristics between patients treated with breast conserving surgery + whole breast irradiation or mastectomy for breast cancer.

Recent observations regarding long-term outcomes among patients with early-stage breast cancer who underwent breast-conserving surgery plus whole-breast irradiation or mastectomy are from a small number of registry-based studies.

Therefore, these findings may overestimate differences in survival between the two groups, compared with randomized controlled trials conducted in the 1980s.

This study performed a propensity score-matched analysis in a cohort of 9710 patients aged <70 years who underwent breast conserving surgery + whole breast irradiation or mastectomy without external radiotherapy for a first primary breast cancer (pT1-2, N0-3a) at the European Institute of Oncology between 2000 and 2008.

Patients were matched by propensity score.

ELIGIBILITY:
Inclusion Criteria:

* First primary breast cancer
* pT1-2
* pN0-3a
* Surgery performed at European Institute of Oncology between 2000 and 2008

Exclusion Criteria:

* pT>=3
* Neoadjuvant treatment
* Presence of metastatic breast disease at the time of admission or within 3 months

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospectively analysis of patients who received treatment for invasive breast cancer at the European Institute of Oncology between January 1, 2000, and December 31, 2008.
  The original cohort comprised 9710 eligible patients with breast cancer, of whom 2289 (23.6%) underwent breast conserving surgery + whole breast irradiation and 7421 (76.4%) underwent mastectomy alone.
  After propensity score matching, 1970 of the 2289 patients who underwent mastectomy (86.1%) were successfully matched to 1970 patients who underwent breast conserving surgery.
Sampling Method: Non-Probability Sample
Enrollment: 9710 (Actual)
Dates: Start 2000-01 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of ipsilateral breast tumor recurrence | 10 years
  Incidence of ipsilateral breast tumor recurrence in breast conserving surgery group compared to mastectomy group
Cumulative incidence of axillary lymph node recurrence | 10 years
  cumulative incidence of axillary lymph node recurrence in breast conserving surgery group compared to mastectomy group
Cumulative incidence of contralateral breast cancer | 10 years
  Cumulative incidence of contralateral breast cancer in breast conserving surgery group compared to mastectomy group
Rate of distant metastasis | 10 years
  Incidence of distant metastasis in breast conserving surgery group compared to mastectomy group
Cumulative incidence of breast cancer specific survival | 10 years
  Cumulative incidence of breast cancer specific survival in breast conserving surgery group compared to mastectomy group
Rate of overall survival | 10 years
  Incidence of survival in breast conserving surgery group compared to mastectomy group

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Magnoni, MD, Principal Investigator — European Institute of Oncology

IPD SHARING:
Plan to Share IPD: No